CLINICAL TRIAL: NCT01218321
Title: Phase 1 Study for Measuring the Effect of Antiepileptic Drugs on Mitochondrial Activity
Brief Title: The Effect of Anti-epileptic Drugs on Mitochondrial Activity
Status: Completed | Type: Observational
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Sponsor
Other Study IDs: 0582-09-HMO-CTIL
Record Dates: First submitted 2010-10-07; First posted 2010-10-11 (Estimated); Last update posted 2018-03-06 (Actual); Status verified 2010-10

CONDITIONS: Epilepsy
Keywords: antiepileptic drugs; mitochondria
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — White blood cells from peripheral blood samples
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Antiepileptic treatment group: Group of patients treated by antiepileptic medications
  Interventions: Biological: antiepileptic treatment

INTERVENTIONS:
Biological: antiepileptic treatment — White blood cells from peripheral blood samples
  Other Names: study group

SUMMARY:
This study is based on the hypothesis that antiepileptic drugs (other than Valproic acid) have an effect on the mitochondrial oxidative phosphorylation.

The objective of this study is to evaluate this effect in an accessible tissue-human peripheral white blood cells.

DETAILED DESCRIPTION:
Antiepileptic drugs adverse reactions, including hepatotoxicity, are rare but potentially fatal, especially among children. Although the mechanism of the liver toxicity remains elusive, mitochondrial oxidative stress, has been hypothesized to play a role.

Most of the studies addressing antiepileptic drug effects on the mitochondria discuss the effect of valproic acid. The exact mechanisms involved in the drug-induced effects on oxidative phosphorylation are still far from being resolved. Most of the studies investigated the effect of valproic acid by using animal models or different in vitro methods.Mitochondrial diseases should be considered as a risk factor for valproic acid-induced hepatotoxicity, and there is a consensus for avoiding the administration of the drug for these patientsIs it possible that other antiepileptic drugs have similar effects? The knowledge regarding the effects of other antiepileptic drugs on the mitochondria is relatively scarce.

ELIGIBILITY:
Inclusion Criteria:

* Children between the ages of 3 and 18 years old, who suffer from new onset epilepsy as diagnosed by a certified pediatric neurologist, who do not suffer from a ''metabolic'' disorder, are treated by a single antiepileptic drug, and are not receiving any other type of medication on a chronic basis were included

Exclusion Criteria:

* Children younger than 3 years of age or older than 18 years of age, children who were suspected or known to suffer from a ''metabolic'' disorder or liver dysfunction, children who were under treatment, by any medication on a chronic basis, at the time of the study were excluded.

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children, ages 3 to 18 years old who start new antiepileptic drug treatment for the first time for new onset epilepsy
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2011-01 (Actual); Primary Completion 2011-12 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Itai Berger, MD, Principal Investigator — Hadassah Medical Organization
Locations (1):
- Hadassah-Hebrew University Medical Center, Jerusalem, Israel

REFERENCES:
- [Background] Berger I, Segal I, Shmueli D, Saada A. The effect of antiepileptic drugs on mitochondrial activity: a pilot study. J Child Neurol. 2010 May;25(5):541-5. doi: 10.1177/0883073809352888. PMID 20413803